CLINICAL TRIAL: NCT02999815
Title: Intrathecal Immunoglobulin for Treatment of Adult Patients With Tetanus: a Randomized Controlled 2x2 Factorial Trial
Brief Title: Intrathecal Tetanus Immunoglobulin to Treat Tetanus
Acronym: ITITTT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 03TS
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Tetanus
Keywords: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human tetanus immunoglobulin (Active Comparator): Human tetanus immunoglobulin (Tetagam-P): Injection (prefilled syringe) 250 IU in 1 ml - Intrathecal 500 IU
  Interventions: Procedure: Human tetanus immunoglobulin
- Intramuscular antitoxin (Sham Comparator): Human tetanus immunoglobulin (Tetagam-P): Injection (prefilled syringe) 250 IU in 1 ml - Intramuscular 3000 IU OR Equine antiserum - 21,000 units
  Interventions: Procedure: Human tetanus immunoglobulin; Procedure: Intramuscular antitoxin

INTERVENTIONS:
Procedure: Human tetanus immunoglobulin — Adults admitted to ICU at Hospital for Tropical Diseases will be randomized to receive either human (3000 IU) or equine (21,000 units) intramuscular antitoxin. Second, participants will be randomized to receive the addition of 500 IU intrathecal human antitoxin.
  Other Names: Human tetanus immunoglobulin (Tetagam-P)
Procedure: Intramuscular antitoxin — First, adults admitted to ICU at Hospital for Tropical Diseases will be randomized to receive either human (3000 IU) or equine (21,000 units) intramuscular antitoxin including a 0.05ml test dose (ie 75 units equine antitoxin or 12.5 IU human antitoxin). Second, participants will be randomized with sham procedure
  Arms: Intramuscular antitoxin

SUMMARY:
To establish whether the addition of intrathecal tetanus antitoxin reduces the need for mechanical ventilation in patients with tetanus

DETAILED DESCRIPTION:
The investigators will conduct a randomised partially-blinded controlled 2x2 factorial trial. First, adults admitted to the Intensive Care Unit at the Hospital for Tropical Diseases Ho Chi Minh City will be randomized to receive either human (3000 IU) or equine (21,000 units) intramuscular antitoxin. Second, participants will be randomized to receive either standard treatment with intramuscular antitoxin alone or with the addition of 500 IU intrathecal human antitoxin. Patients with prior antitoxin treatment and those with contra-indications to lumbar puncture or antitoxin treatment will be excluded.

All patients will receive other standard tetanus treatment as deemed necessary by the attending physicians. Spasms will be treated with benzodiazepines as first-line therapy. Patients with spasms not controlled with benzodiazepines will receive tracheostomy, paralysis, magnesium sulphate and mechanical ventilation. Heart rate, BP, temperature and daily drug use will be recorded throughout the ICU stay. Patients will be followed following discharge from hospital until 240 days for disability/ death.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥16 years old) with a clinical diagnosis of generalized tetanus admitted to the intensive care unit (ICU) at the Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

Exclusion Criteria:

* Prior administration of antitoxin during this episode
* Contra-indication to use of human or equine antitoxin
* Contra-indication to lumbar puncture
* Already receiving mechanical ventilation or expected to require this before intrathecal injection can be given
* Pregnancy
* Informed consent not obtained

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Requirement for mechanical ventilation during ICU stay | During ICU stay, an average of 3 weeks
  Criteria for mechanical ventilation are oxygen saturation (SpO2) <90%; or partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) <250; or excessive spasms necessitating muscle paralysis.
  These criteria are intended as a guide and the final decision to ventilate a patient rests with the individual doctor responsible for the patient.

SECONDARY OUTCOMES:
Duration of ICU stay | During ICU stay, an average of 3 weeks
Duration of hospital stay | During hospital stay, an average of 5 weeks
Duration of mechanical ventilation | During hospital stay, an average of 5 weeks
In hospital and 240 day mortality | 240 days
In hospital and 240 day disability | 240 days
New antibiotic prescription during ICU stay | During ICU stay, an average of 3 weeks
  New antibiotic prescription during ICU stay (excluding antibiotics for tetanus or initial entry site infection)
Incidence of Ventilator Associated Pneumonia | During hospital stay, an average of 5 weeks
  Definition of Ventilator associated pneumonia (VAP):
  Mechanical ventilation for at least 48 hours and with the tube in place within the last 48 hours and 2 of:
  * Temperature > 38°C or < 36°C
  * White blood cell count <4.0 x 109/L or ≥12 x 109/L
  * Purulent respiratory secretions
  * New or progressive changes on chest radiography (for VAP) Plus for microbiologically confirmed VAP
  * Bacterial growth of ≥105 cfu/ml from endotracheal aspirate (ETA) (or ≥104 cfu/ml from Broncho Alveolar Lavage (BAL))
Incidence of clinical syndrome of autonomic nervous system dysfunction | 240 days
  At least 3 of the following criteria:
  * Tachycardia Heart Rate (HR)> 100 bpm
  * Hypertension Systolic Blood Pressure (SBP) > 140 mmHg
  * Hypotension Mean Arterial Pressure (MAP) < 60 mmHg
  * Pyrexia > 38°C
  * Alteration between hypertension and hypotension
Total dose of benzodiazepines and pipecuronium during hospital stay | During hospital stay, an average of 5 weeks
Incidence of adverse events | During hospital stay, an average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minh Yen Lam, MD, Principal Investigator — Oxford University Clinical Research Unit
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang D, Pu X, Wu J, Li M, Liu P. Rapid, sensitive, and specific detection of Clostridium tetani by loop-mediated isothermal amplification assay. J Microbiol Biotechnol. 2013 Jan;23(1):1-6. doi: 10.4014/jmb.1205.05063. PMID 23314360
- [Background] Thwaites CL, Yen LM, Nga NT, Parry J, Binh NT, Loan HT, Thuy TT, Bethell D, Parry CM, White NJ, Day NP, Farrar JJ. Impact of improved vaccination programme and intensive care facilities on incidence and outcome of tetanus in southern Vietnam, 1993-2002. Trans R Soc Trop Med Hyg. 2004 Nov;98(11):671-7. doi: 10.1016/j.trstmh.2004.01.008. PMID 15363647
- [Background] Rosenthal VD, Maki DG, Salomao R, Moreno CA, Mehta Y, Higuera F, Cuellar LE, Arikan OA, Abouqal R, Leblebicioglu H; International Nosocomial Infection Control Consortium. Device-associated nosocomial infections in 55 intensive care units of 8 developing countries. Ann Intern Med. 2006 Oct 17;145(8):582-91. doi: 10.7326/0003-4819-145-8-200610170-00007. PMID 17043340
- [Background] Thwaites CL, Yen LM, Loan HT, Thuy TT, Thwaites GE, Stepniewska K, Soni N, White NJ, Farrar JJ. Magnesium sulphate for treatment of severe tetanus: a randomised controlled trial. Lancet. 2006 Oct 21;368(9545):1436-43. doi: 10.1016/S0140-6736(06)69444-0. PMID 17055945
- [Background] Ildirim I. A new treatment for neonatal tetanus. Antitetanic serum and prednisolone given together intrathecally. Turk J Pediatr. 1967 Jul;9(3):89-95. No abstract available. PMID 5630851
- [Background] St-Amour I, Pare I, Alata W, Coulombe K, Ringuette-Goulet C, Drouin-Ouellet J, Vandal M, Soulet D, Bazin R, Calon F. Brain bioavailability of human intravenous immunoglobulin and its transport through the murine blood-brain barrier. J Cereb Blood Flow Metab. 2013 Dec;33(12):1983-92. doi: 10.1038/jcbfm.2013.160. Epub 2013 Sep 18. PMID 24045402
- [Background] Miana-Mena FJ, Roux S, Benichou JC, Osta R, Brulet P. Neuronal activity-dependent membrane traffic at the neuromuscular junction. Proc Natl Acad Sci U S A. 2002 Mar 5;99(5):3234-9. doi: 10.1073/pnas.052023599. PMID 11880654
- [Background] Sancho A, Melchiorri D, Abadie E; Committee for Medicinal Products for Human Use, European Medicines Agency. More on influenza vaccine in young children. N Engl J Med. 2012 Jun 28;366(26):2528; author reply 2528-9. doi: 10.1056/NEJMc1205643. No abstract available. PMID 22738111
- [Background] Lalli G, Schiavo G. Analysis of retrograde transport in motor neurons reveals common endocytic carriers for tetanus toxin and neurotrophin receptor p75NTR. J Cell Biol. 2002 Jan 21;156(2):233-9. doi: 10.1083/jcb.200106142. Epub 2002 Jan 21. PMID 11807088
- [Background] FRIEDEMANN U, TRAUB FB. Pathogenesis of local tetanus in the dog and the cat. J Immunol. 1949 Sep;63(1):23-8. No abstract available. PMID 18139406
- [Background] Roux E, Borrel A. Tetanos Cerebral et immunite contre le tetanus. Ann Inst Pasteur (Paris) [Internet]. 1898;12(4):525-35. Available from: https://archive.org/stream/annalesdelinstit12inst
- [Background] Florey H, Fildes P. Tetanus . -Vii . the Treatment of Tetanus in Rabbits By Large Intrathecal Doses of Antitoxin . Br J Exp Pathol. 1927;(October):393-7
- [Background] Sherrington BYCS. The serum treatment of experimental tetanus in monkeys. Lancet. 1917;964:54-68
- [Background] Sedaghatian MR. Intrathecal serotherapy in neonatal tetanus: a controlled trial. Arch Dis Child. 1979 Aug;54(8):623-5. doi: 10.1136/adc.54.8.623. PMID 389175
- [Background] Ildirim I. Intrathecal serotherapy of tetanus. I. Explanation of complications. II. Comparison of intrathecal tetanus immune globulin and tetanus antitoxin. Turk J Pediatr. 1974 Jul;16(3):103-10. No abstract available. PMID 4480716
- [Background] Miranda-Filho Dde B, Ximenes RA, Barone AA, Vaz VL, Vieira AG, Albuquerque VM. Randomised controlled trial of tetanus treatment with antitetanus immunoglobulin by the intrathecal or intramuscular route. BMJ. 2004 Mar 13;328(7440):615. doi: 10.1136/bmj.38027.560347.7C. Epub 2004 Mar 5. PMID 15003976
- [Background] Wateba M, Diop S, Nichols S, Patassi A, Adjo S, Gbadamassi G, Tidjani O. [Intrathecal therapy with 1 500 UI of antitetanic serum and 1.5 g of intravenous metronidazole: prognosis of tetanus in hospitalized patients in Togo]. Sante. 2008 Jul-Sep;18(3):125-9. doi: 10.1684/san.2008.0115. French. PMID 19359232
- [Background] Menon J, Mathews L. Intrathecal immunoglobulin in the treatment of tetanus. Indian Pediatr. 2002 Jul;39(7):654-7. No abstract available. PMID 12147891
- [Background] Sun KO, Chan YW, Cheung RT, So PC, Yu YL, Li PC. Management of tetanus: a review of 18 cases. J R Soc Med. 1994 Mar;87(3):135-7. doi: 10.1177/014107689408700306. PMID 8158589
- [Background] Abrutyn E, Berlin JA. Intrathecal therapy in tetanus. A meta-analysis. JAMA. 1991 Oct 23-30;266(16):2262-7. PMID 1833565
- [Background] Kabura L, Ilibagiza D, Menten J, Van den Ende J. Intrathecal vs. intramuscular administration of human antitetanus immunoglobulin or equine tetanus antitoxin in the treatment of tetanus: a meta-analysis. Trop Med Int Health. 2006 Jul;11(7):1075-81. doi: 10.1111/j.1365-3156.2006.01659.x. PMID 16827708
- [Background] Agarwal M, Thomas K, Peter JV, Jeyaseelan L, Cherian AM. A randomized double-blind sham-controlled study of intrathecal human anti-tetanus immunoglobulin in the management of tetanus. Natl Med J India. 1998 Sep-Oct;11(5):209-12. PMID 10997166
- [Background] Rodrigo C, Fernando D, Rajapakse S. Pharmacological management of tetanus: an evidence-based review. Crit Care. 2014 Mar 26;18(2):217. doi: 10.1186/cc13797. PMID 25029486
- [Background] Govindaraj GM, Riyaz A. Current practice in the management of tetanus. Crit Care. 2014 May 27;18(3):145. doi: 10.1186/cc13894. PMID 25042788
- [Background] Health Protection Agency. HPA expert working group interim guidance on the use of tetanus immunoglobulin for the treatment of Tetanus [Internet]. 2013. Available from: https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/400084/expert_working_group_interim_guidance_on_the_use_of_tetanus_immunoglobulin_for_the_treatment_of_Tetanus.pdf
- [Background] NATION NS, PIERCE NF, ADLER SJ, CHINNOCK RF, WEHRLE PF. Tetanus; the use of human hyperimmune globulin in treatment. Calif Med. 1963 Jun;98(6):305-7. PMID 13937706
- [Background] Naguwa SM, Nelson BL. Human serum sickness. Clin Rev Allergy. 1985 Feb;3(1):117-26. doi: 10.1007/BF02993045. No abstract available. PMID 3884125
- [Background] McCracken GH Jr, Dowell DL, Marshall FN. Double-blind trial of equine antitoxin and human immune globulin in tetanus neonatorum. Lancet. 1971 Jun 5;1(7710):1146-9. doi: 10.1016/s0140-6736(71)91659-x. No abstract available. PMID 4102858
- [Background] Smith JW, Schallibaum EM. The therapeutic effect of homologous and heterologous antitoxins in experimental diphtheria and tetanus. Br J Exp Pathol. 1970 Feb;51(1):73-80. PMID 4985287
- [Background] Calvo AC, Olivan S, Manzano R, Zaragoza P, Aguilera J, Osta R. Fragment C of tetanus toxin: new insights into its neuronal signaling pathway. Int J Mol Sci. 2012;13(6):6883-6901. doi: 10.3390/ijms13066883. Epub 2012 Jun 7. PMID 22837670
- [Background] Health Protection Agency. Tetanus [Internet]. Information for Health Professionals. 2013. Available from: http://www.hpa.org.uk/webc/HPAwebFile/HPAweb_C/1194947374762
- [Background] Sanders RK, Martyn B, Joseph R, Peacock ML. Intrathecal antitetanus serum (horse) in the treatment of tetanus. Lancet. 1977 May 7;1(8019):974-7. doi: 10.1016/s0140-6736(77)92278-4. PMID 67468
- [Background] Smith JW. Intracerebral antitoxin in experimental tetanus. Br J Exp Pathol. 1966 Feb;47(1):17-24. No abstract available. PMID 5908697
- [Background] Loan HT, Parry J, Nga NT, Yen LM, Binh NT, Thuy TT, Duong NM, Campbell JI, Thwaites L, Farrar JJ, Parry CM. Semi-recumbent body position fails to prevent healthcare-associated pneumonia in Vietnamese patients with severe tetanus. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):90-7. doi: 10.1016/j.trstmh.2011.10.010. Epub 2011 Dec 22. PMID 22197012
- [Background] Thwaites CL, Yen LM, Glover C, Tuan PQ, Nga NT, Parry J, Loan HT, Bethell D, Day NP, White NJ, Soni N, Farrar JJ. Predicting the clinical outcome of tetanus: the tetanus severity score. Trop Med Int Health. 2006 Mar;11(3):279-87. doi: 10.1111/j.1365-3156.2006.01562.x. PMID 16553907
- [Background] Luangasanatip N, Hongsuwan M, Lubell Y, Limmathurotsakul D, Teparrukkul P, Chaowarat S, Day NP, Graves N, Cooper BS. Long-term survival after intensive care unit discharge in Thailand: a retrospective study. Crit Care. 2013 Oct 3;17(5):R219. doi: 10.1186/cc13036. PMID 24090280
- [Background] Mchil Ugwu GI. Neonatal Tetanus in Varri Niger Delta: A Ten Year Retrospective Study. CJMedRes. 2010;4:3-7
- [Background] Barlow JL, Mung'Ala-Odera V, Gona J, Newton CR. Brain damage after neonatal tetanus in a rural Kenyan hospital. Trop Med Int Health. 2001 Apr;6(4):305-8. doi: 10.1046/j.1365-3156.2001.00705.x. PMID 11348521
- [Background] Neequaye J, Nkrumah FK. Failure of intrathecal antitetanus serum to improve survival in neonatal tetanus. Arch Dis Child. 1983 Apr;58(4):276-8. doi: 10.1136/adc.58.4.276. PMID 6342543
- [Background] Vakil BJ, Armitage P, Clifford RE, Laurence DR. Therapeutic trial of intracisternal human tetanus immunoglobulin in clinical tetanus. Trans R Soc Trop Med Hyg. 1979;73(5):579-83. doi: 10.1016/0035-9203(79)90058-0. PMID 583378
- [Background] Thwaites CL, Beeching NJ, Newton CR. Maternal and neonatal tetanus. Lancet. 2015 Jan 24;385(9965):362-70. doi: 10.1016/S0140-6736(14)60236-1. Epub 2014 Aug 19. PMID 25149223
- [Background] Robert R, Rouffineau J, Cremault A, Bauple JL, Pourrat O, Gil R, Patte D. [Reversible paraplegia following intrathecal injection of high doses of human gammaglobulins in the treatment of low-grade tetanus. 4 cases]. Presse Med. 1984 Sep 22;13(32):1947-9. French. PMID 6207524
- [Background] Dodou K. Intrathecal route of drug delivery can save lives or improve quality of life [Internet]. Pharmaceutical Journal. 2012. p. 9-12. Available from: http://www.pjonline.com/news/intrathecal_route_of_drug_delivery_can_save_lives_or_improve_quality_of_life
- [Background] Dodou K. Intrathecal route of drug delivery can save lives or improve quality of life. Pharmaceutical Journal. 2012. p. 9-12
- [Background] Munts AG, van der Plas AA, Voormolen JH, Marinus J, Teepe-Twiss IM, Onkenhout W, van Gerven JM, van Hilten JJ. Intrathecal glycine for pain and dystonia in complex regional pain syndrome. Pain. 2009 Nov;146(1-2):199-204. doi: 10.1016/j.pain.2009.07.030. Epub 2009 Aug 14. PMID 19683392
- [Background] Lim ES, Lee IO. Effect of intrathecal glycine and related amino acids on the allodynia and hyperalgesic action of strychnine or bicuculline in mice. Korean J Anesthesiol. 2010 Jan;58(1):76-86. doi: 10.4097/kjae.2010.58.1.76. Epub 2010 Jan 31. PMID 20498816
- [Background] Lee IO, Son JK, Lim ES, Kim YS. Pharmacology of intracisternal or intrathecal glycine, muscimol, and baclofen in strychnine-induced thermal hyperalgesia of mice. J Korean Med Sci. 2011 Oct;26(10):1371-7. doi: 10.3346/jkms.2011.26.10.1371. Epub 2011 Oct 1. PMID 22022192
- [Background] Andrewes F. On the intrathecal route for the administration of tetanus antitoxin. Lancet. 1917;189(May):682-6
- [Background] Gupta PS, Kapoor R, Goyal S, Batra VK, Jain BK. Intrathecal human tetanus immunoglobulin in early tetanus. Lancet. 1980 Aug 30;2(8192):439-40. doi: 10.1016/s0140-6736(80)91883-8. PMID 6106095
- [Background] Ahmad A, Qaisar I, Naeem M, Mazhar AU, Ashfaq M. Intrathecal anti-tetanus human immunoglobulin in the treatment of neonatal tetanus. J Coll Physicians Surg Pak. 2011 Sep;21(9):539-41. PMID 21914410
- [Background] Mongi PS, Mbise RL, Msengi AE, Do Amsi DM. Tetanus neonatorum--experience with intrathecal serotherapy at Muhimbili Medical Centre, Dar es Salaam, Tanzania. Ann Trop Paediatr. 1987 Mar;7(1):27-31. doi: 10.1080/02724936.1987.11748469. PMID 2439000
- [Background] Rowbotham MC. Pain's policy on the spinal administration of drugs. Pain. 2010 Jun;149(3):415-416. doi: 10.1016/j.pain.2010.02.027. Epub 2010 Mar 3. No abstract available. PMID 20202752
- [Background] Eisenach JC, Shafer SL, Yaksh T. The need for a journal policy on intrathecal, epidural, and perineural administration of non-approved drugs. Pain. 2010 Jun;149(3):417-419. doi: 10.1016/j.pain.2010.02.028. Epub 2010 Mar 15. No abstract available. PMID 20227830
- [Background] Geeta MG, Krishnakumar P, Mathews L. Intrathecal tetanus immunoglobulins in the management of tetanus. Indian J Pediatr. 2007 Jan;74(1):43-5. doi: 10.1007/s12098-007-0025-y. PMID 17264452
- [Background] Turillazzi E, Neri M, Pomara C, Riezzo I, Fineschi V. An immunohistochemical study on a tetanus fatal case using toxin fragment C (TTC). Should it be a useful diagnostic tool? Neuropathology. 2009 Feb;29(1):68-71. doi: 10.1111/j.1440-1789.2008.00912.x. Epub 2008 Apr 15. PMID 18422910
- [Derived] Van Hao N, Loan HT, Yen LM, Kestelyn E, Hong DD, Thuy DB, Nguyen NT, Duong HTH, Thuy TTD, Nhat PTH, Khanh PNQ, Dung NTP, Phu NH, Phong NT, Lieu PT, Tuyen PT, Hanh BTB, Nghia HDT, Oanh PKN, Tho PV, Tan Thanh T, Turner HC, van Doorn HR, Van Tan L, Wyncoll D, Day NP, Geskus RB, Thwaites GE, Van Vinh Chau N, Thwaites CL. Human versus equine intramuscular antitoxin, with or without human intrathecal antitoxin, for the treatment of adults with tetanus: a 2 x 2 factorial randomised controlled trial. Lancet Glob Health. 2022 Jun;10(6):e862-e872. doi: 10.1016/S2214-109X(22)00117-6. PMID 35561721
- [Derived] Loan HT, Yen LM, Kestelyn E, Hao NV, Thanh TT, Dung NTP, Turner HC, Geskus RB, Wolbers M, Tan LV, Van Doorn HR, Day NP, Wyncoll D, Hien TT, Thwaites GE, Vinh Chau NV, Thwaites CL. Intrathecal Immunoglobulin for treatment of adult patients with tetanus: A randomized controlled 2x2 factorial trial. Wellcome Open Res. 2018 Nov 5;3:58. doi: 10.12688/wellcomeopenres.14587.2. eCollection 2018. PMID 30809591